CLINICAL TRIAL: NCT00568997
Title: A Prospective 10 Year Observational Registry of Pediatric Subjects (Age Greater Than or Equal to Two Years to Age Less Than or Equal to 17 Years) With Atopic Dermatitis Who Have Used Elidel Cream 1% (Pimecrolimus)
Brief Title: 10 Year Registry of Children (Ages 2-17 Years) With Eczema That Have Used Pimecrolimus
Acronym: PEER
Status: Active, not recruiting | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Clinical Research Computing Unit (University of Pennsylvania) (Other)
Responsible Party: Sponsor
Other Study IDs: CASM981C2311
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis eczema pediatric pimecrolimus malignancy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Single-group Open Label Registry of patients exposed to Elidel/Pimecrolimus
  Interventions: Drug: Pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus 1% cream
  Other Names: Elidel

SUMMARY:
This study will examine the risk of systemic malignancies in pediatric patients with atopic dermatitis exposed to Elidel 1% cream.

DETAILED DESCRIPTION:
Registry study to examine the risk of systemic malignancies in pediatric patients with atopic dermatitis exposed to Elidel 1% cream.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* greater than or equal to 2 years and less than or equal to 17 years at enrollment
* diagnosis of atopic dermatitis (confirmed by treating physician)
* applied pimecrolimus cream 1 % 6 weeks out of past 24 weeks

Exclusion Criteria:

* past or present history of systemic malignancy, skin malignancy, or lymphoproliferative disease
* past or present use of oral immunosuppressive therapy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (ages 2-17 years)
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2005-06-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of systemic malignancies in pediatric subjects with atopic dermatitis who have been exposed to pimecrolimus 1% cream | 10 years of observation with 6-month reporting intervals

SECONDARY OUTCOMES:
The incidence rate of lymphoma in pediatric subjects with atopic dermatitis who have been exposed to pimecrolimus 1% cream | 10 years of observation with 6-month reporting intervals
The incidence rate of thyroid cancer in pediatric subjects with atopic dermatitis who have been exposed to pimecrolimus 1% cream | 10 years of observation with 6-month reporting intervals
The incidence rate of cutaneous malignancy in pediatric subjects with atopic dermatitis who have been exposed to pimecrolimus 1% cream | 10 years of observation with 6-month reporting intervals

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health
Locations (1):
- Registry, Philadelphia, Pennsylvania, United States